CLINICAL TRIAL: NCT05314205
Title: Long-term Outcome of Ligation of Inter-sphincteric Fistula Tract (LIFT) for Management of Trans-sphincteric Anal Fistula
Brief Title: Ligation of Inter-sphincteric Fistula Tract for Management of Anal Fistula
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdulkarim Hasan, Laboratory coordinator, Al-Azhar University
Other Study IDs: AUHS2101201
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ligation of inter-sphincteric fistula tract — The surgical treatment was achieved through identification of the fistula by injecting hydrogen peroxide (H2O2) through the external opening. Probing of the fistulous tract by a metallic probe for proper identification of the fistula in the inter-sphincteric plane.
  Perpendicular skin incision (about 1 cm) was done at inter-sphinctric zone, perpendicular to the fistulous tract. Dissection between the internal and external sphincters and identification of the fistula.
  Finally, Ligation and transection of the tract in inter-sphinctric space followed by excision of a segment and transferred for histopathology examination. Trans-fixation suture was applied near to the internal mucosal opening of the divided tract to confirm closure using polyglactin suture 2/0. Insertion of a probe to check the closure of the tract segments.
  The remaining part of the tract was curetted till external opening and left for spontaneous healing.

SUMMARY:
After abscess formation, an anal fistula is a common consequence, with crypto-glandular infection being the most commonly accepted causative cause. The goal of this study was to see how well closure of the inter-sphincteric fistula tract affects the outcome of trans-sphincteric fistula surgery. Patients with perianal trans-sphincteric fistulas who underwent ligation were studied prospectively. All patients had the identical anesthetic approach, followed by the operation with two years' follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with trans-sphincteric peri-anal fistulas (according to magnetic resonance fistulogram) of crypto-glandular source with no previous fistula surgery

Exclusion Criteria:

* Individuals with recurrent fistulae or had specific pathology, like Crohn's disease.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from surgery clinic at AlAzhar Hospital
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Post-operative complication | 2 years
  The post-operative follow-up was done in an outpatient setting, with weekly visits for the first month, every two months for six months and then by phone calls to know recurrence and infection occurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Abdulkarim Hasan, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided